CLINICAL TRIAL: NCT07149584
Title: Erector Spinae Plane Block Versus Thoracic Paravertebral Block in Laparoscopic Cholecystectomy: A Randomized Controlled Trial on Opioid Consumption
Brief Title: Erector Spinae Plane Block Versus Thoracic Paravertebral Block in Laparoscopic Cholecystectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Ozlem Turhan, Attending Anesthesiologist, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2025/1127
Record Dates: First submitted 2025-08-23; First posted 2025-09-02 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Pain, Acute Postoperative
Keywords: postoperative pain; erector spinal plane block; thoracic paravertebral block
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1: ESPB (Experimental): Erector spinal plane block
  Interventions: Procedure: ESPB
- Group 2: TPVB (Experimental): Thoracic paravertebral block
  Interventions: Procedure: TPVB
- Group 3: IV (Experimental): intravenous analgesia
  Interventions: Procedure: IV

INTERVENTIONS:
Procedure: ESPB — 10 mL of 0.375% bupivacaine is injected on each side between the deep fascia of the erector spinae muscle and the transverse process. Additionally, tramadol is administered via intravenous patient-controlled analgesia.
  Arms: Group 1: ESPB
Procedure: TPVB — 10 mL of 0.375% bupivacaine is injected on each side between the superior costotransverse ligament and the pleura.
  Arms: Group 2: TPVB
Procedure: IV — Tramadol is administered via intravenous patient-controlled analgesia.
  Arms: Group 3: IV

SUMMARY:
The study is planned as a single-center prospective randomized study and includes patients undergoing laparoscopic cholecystectomy. The aim of this study is to compare postoperative analgesic efficacy of erector spinae plane block and thoracic paravertebral block. Primary outcome is 24-hour postoperative opioid consumption.

DETAILED DESCRIPTION:
All patients in the operating room receive the same anesthetic management under standard monitoring modalities. Both erector spinae plane block (ESPB) and thoracic paravertebral block (TPVB) are performed under ultrasound guidance at the T8 level using a linear probe and a longitudinal out-of-plane technique before induction of anesthesia. For ESPB, 10 mL of 0.375% bupivacaine is injected bilaterally between the deep fascia of the erector spinae muscle and the transverse process. For TPVB, 10 mL of 0.375% bupivacaine is injected bilaterally into the paravertebral space. After standard anesthesia induction, anesthesia is maintained with inhalation agents. Four milligrams of dexamethasone and 8 mg of ondansetron are administered for postoperative nausea and vomiting prophylaxis. As part of multimodal analgesia, all patients receive 1 g of paracetamol and 20 mg of tenoxicam.

All patients are followed according to a standardized postoperative analgesia protocol, which includes tramadol patient-controlled analgesia (10 mg bolus, 20-minute lockout). Postoperative static and dynamic pain scores are evaluated using the numeric rating scale (NRS) at 0, 1, 4, 6, 12, 18, and 24 hours. If the NRS score is greater than 3, 0.5 mg/kg meperidine is administered as rescue analgesia.

ELIGIBILITY:
Inclusion Criteria:

* Elective cholecystectomy
* Age >18years
* American Society of Anesthesiologists classification I-III

Exclusion Criteria:

* Presence of contraindications for using regional anesthesia ( not having patient approval, bleeding diathesis or use of anticoagulants, infection at the injection site, and allergy to local anesthetics)
* Chronic analgesic use
* Open cholecystectomy or conversion to open cholecystectomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Tramadol consumption | postoperative 24 hours
  amount of postoperative 24-hour tramadol consumption

SECONDARY OUTCOMES:
Amount of fentanyl | during surgery
  Amount of fentanyl used intraoperatively
Static and dynamic pain score | postoperative 24 hours
  Static and dynamic pain scores are assessed with numeric rating scale at 0., 1., 4., 6., 12., 18. and 24. hours.
First rescue analgesic time | postoperative 24 hours
  The first time patient required rescue analgesic.
Number of patients required rescue analgesic. | postoperative 24 hours
  If the NRS score is greater than 3, 0.5 mg/kg meperidine is administered as rescue analgesia.
Nausea and vomiting | postoperative 24 hours
  Number of patients experienced postoperative nausea and vomiting
Complications | postoperative 24 hours
  Number of patients experienced complications postoperatively
Quality of recovery | postoperative 24 hours
  Patient recovery quality is evaluated using the Quality of Recovery-15 (QoR-15) questionnaire. QoR-15 scores range from 0 (extremely poor quality of recovery) to 150 (excellent quality of recovery).
Length of hospital stay | up to 1 week
  Length of hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Özlem Turhan, Principal Investigator — Istanbul Faculty of Medicine
Locations (1):
- Istanbul University, Istanbul Faculty of Medicine, Istanbul, Turkey (Türkiye)